CLINICAL TRIAL: NCT00808873
Title: A Randomized Control Trial of a Socio-Educational Intervention for Rural Suicide Attempters in Tianjin Municipality and Shandong Province of China
Brief Title: Socio-Educational Intervention for Rural Suicide Attempters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing HuiLongGuan Hospital (Other)
Collaborators: Suicide Prevention International (Other); Harvard University (Other); University of Rochester (Other); People's Hospital of Yuncheng County (Unknown); Bureau of Health of Ji County (Unknown)
Responsible Party: Xianyun Li, Beijing Hui Long Guan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2008-7
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-11

CONDITIONS: Suicide, Attempted
Keywords: attempted suicide; socio-educational intervention; follow up study
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): brief education and 6 follow-up visits
  Interventions: Other: socio-educational intervention
- 2 (No Intervention): treatment-as-usual

INTERVENTIONS:
Other: socio-educational intervention — brief mental health education and 6 follow-up visits
  Other Names: psychosocial intervention on suicide prevention
  Arms: 1

SUMMARY:
Compared to a treatment-as-usual group, providing brief mental health education to suicide attempters from rural parts of China at the time of their treatment in the emergency departments of general hospitals or local clinics and 6 home-visits (FOR those subjects WITH PHONES refuse home visits, THE INTERVIEWS WILL BE CONDUCTED OVER THE PHONE) over the twelve months after the attempt demonstrate continuing concern about the attempters ('befriending'), strengthen their social support networks and improve their problem-solving skills will significantly reduce their hopelessness, the severity of depressive symptoms, and level of suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* suicide attempters
* must be 18 years or older
* no-zero intent to die

Exclusion Criteria:

* with communication difficulties
* living outside of the research sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-02 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
the severity of depressive symptoms | one year

SECONDARY OUTCOMES:
frequency and intensity of suicidal ideation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Xianyun Li, Bachelor, Master of Medicine, Principal Investigator — Beijing HuiLongGuan Hospital
Locations (1):
- People's Hospital of Yuncheng County, Yuncheng County, Shandong, China